CLINICAL TRIAL: NCT02954120
Title: Evaluation Of Lipid Peroxidation, Oxidative DNA Damage And Total Antioxidant Status In Patients With Periodontitis And Polycystic Ovary Syndrome: A Cross Sectional Study
Brief Title: Chronic Periodontitis and Polycystic Ovary Syndrome
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: PCOSandCP
Record Dates: First submitted 2016-10-28; First posted 2016-11-03 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Polycystic Ovary Syndrome; Chronic Periodontitis
Keywords: 8- hydroxy -2´- deoxyguanosine; Malondialdehyde; Total antioxidant status; Oxidative stres
MeSH Terms: conditions — Polycystic Ovary Syndrome; Chronic Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Serum and saliva samples were obtained and stored until biochemical analyses
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- (PCOS-CP-): systemically and periodontally healthy participants
  Interventions: Other: no intervention provided
- (PCOS-CP+): systemically healthy participants with CP
  Interventions: Other: no intervention provided
- (PCOS+CP-): PCOS participants with periodontally healthy
  Interventions: Other: no intervention provided
- (PCOS+CP+): PCOS participants with CP
  Interventions: Other: no intervention provided

INTERVENTIONS:
Other: no intervention provided

SUMMARY:
Background: The aim of this study was to investigate the levels of malondialdehyde (MDA), total antioxidant status (TAS), 8-hydroxy-2´- deoxyguanosine (8-OHdG) in blood serum and saliva samples in female patients with chronic periodontitis (CP) and to compared healthy individuals.

Materials and Methods: A total of 88 women were into four groups each which were consisted of twenty-two subjects. Groups were designed as periodontally and systemically healthy women (PCOS-CP-); periodontally healthy women with polycystic ovary syndrome (PCOS) (PCOS+CP-), systemically healthy women with CP (PCOS-,CP+) and women with PCOS and CP (PCOS+CP+). Serum and salivary samples were obtained, clinical periodontal parameters were recorded. MDA, TAS, 8-OHdG levels were measured as biochemically.

DETAILED DESCRIPTION:
RESULTS:

Salivary 8-OHdG levels in the PCOSCP and CP groups were statistically higher than those in both the PCOSPH and the PH groups (P < 0.05). There was no statistical difference between the PCOSCP, CP, and PCOSPH groups with regard to salivary MDA and TAS levels (P > 0.05). Highest serum 8-OHdG and MDA levels and lowest serum TAS levels were seen in the PCOSCP group (P < 0.05). Serum 8-OHdG and MDA levels in the PCOSPH group were higher than those in both systemically healthy groups (PH and CP) (P < 0.05). Salivary TAS levels were highest (P < 0.05) in the PH group. There was no statistical difference between the CP and PCOSPH groups, but serum TAS levels were lower than those in the PH group (P < 0.05).

CONCLUSIONS:

CP, which led to an increase in serum and salivary 8-OHdG and MDA levels and a decrease in serum TAS levels in patients with PCOS, contributed to increased OS. This effect was more prominent in serum levels than in salivary levels.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed non-obese PCOS patients
* Never smokers
* Had no history of systemic disease
* BMI<25 kg/m2
* Participants had ≥20 teeth present.

Exclusion Criteria:

* Pregnancy
* Lactation
* Hemoglobin A1c (HbA1c) ≥ 6.5%
* 2-h oral glucose tolerance test (OGTT-2h) ≥200
* Cushing syndrome, non-classic congenital adrenal hyperplasia, hyperprolactinemia, thyroid dysfunction, and androgen-secreting tumors
* Any drug use within the past 6 months
* Periodontal treatment within the past 6 months

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All participants were recruited among women at the Department of Obstetrics and Gynecology, School of Medicine, Ataturk University
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2013-05; Primary Completion 2015-05 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
8-OHdG levels (nanogram per mililiter(ng/mL)) | appoximately 2 years
  by ELISA test
MDA levels (micromole per liter (µmol/L)) | appoximately 2 years
  by ELISA test
TAS levels (millimolar per liter (mmol /L)) | appoximately 2 years
  by ELISA test
Plaque Index (PI) | appoximately 2 years
  Silnes-Löe Periodondal İndex
Gingival Index (GI) | appoximately 2 years
  Löe-Silness Periodontal Index
Bleeding on probing (BOP) | appoximately 2 years
  Gİngival Bleeding Index
Clinical attachment level (CAL) | Patients were seen one time
  by measuring the distance between the cementoenamel junction and the periodontal pocket base
Probing pocket depth (PD)) | appoximately 2 years
  distance between free gingival margin and periodontal pocket base by usin periodontal probe

SECONDARY OUTCOMES:
number of individuals with chronic periodontitis | appoximately 2 years
  individuals in the group
numberer of individuals with polycystic ovary syndrome | appoximately 2 years
  individuals in the group

CONTACTS AND LOCATIONS:
Overall Officials: Nesrin Saruhan, PhD, Principal Investigator — Eskisehir Osmangazi Üniversitesi; Cenk Fatih Çanakcı, Prof, Study Director — Ataturk University; Saime Ozbek Sebin, Dr, Principal Investigator — Ataturk University; Humeyra Canakcı, Dr, Principal Investigator — Buhara Hastanesi; Metin İngeç, Prof, Principal Investigator — Ataturk University; Ufuk Sezer, Phd, Principal Investigator — Özel Klinik; Ebru Saglam, PhD, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Department of Periodontics, Faculty of Dentistry, Bezmialem Vakif University, Istanbul, Fatih, Turkey (Türkiye)